CLINICAL TRIAL: NCT01837784
Title: Value of Non-invasively Measured Arterial Stiffness and Central Hemodynamics for Guiding Antihypertensive Treatment in Selected Patient Populations
Brief Title: Central Hemodynamics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Prof. Paul Erne, Head of Department of Cardiology, Luzerner Kantonsspital
Other Study IDs: 13024
Record Dates: First submitted 2013-04-16; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Elderly patients
  Interventions: Other: Optimization of blood pressure according to guidelines
- Patients with diabetes mellitus
  Interventions: Other: Optimization of blood pressure according to guidelines
- Patients with heart failure
  Interventions: Other: Optimization of blood pressure according to guidelines
- Patients with resistant hypertension
  Interventions: Other: Optimization of blood pressure according to guidelines

INTERVENTIONS:
Other: Optimization of blood pressure according to guidelines — There is no specific recommendation for the intervention. The goal of the intervention is an optimization of blood pressure control. The intervention is at the discretion of the physician, but should adhere to guidelines. The intervention may therefore embrace measures such as drug prescriptions or lifestyle interventions.

SUMMARY:
Guidelines recommend measuring end organ damage and in particular arterial stiffness in patients with hypertension. However, until now it was not possible to measure arterial stiffness with the use of simple methods. Recently, novel and innovative devices offering determination of arterial stiffness and central hemodynamics from simple and non-invasive arm cuff measurements have now become available. This study therefore evaluates the value of non-invasively measured arterial stiffness and central hemodynamics for guiding antihypertensive treatment in selected patient populations (i.e. elderly patients, patients with diabetes mellitus, patients with heart failure, and patients with resistant hypertension).

ELIGIBILITY:
Inclusion Criteria:

* Patients >70 years (elderly cohort)
* Patients with diabetes mellitus (diabetes cohort)
* Patients with heart failure (heart failure cohort)
* Patients with resistant hypertension (resistant hypertension cohort)

Exclusion Criteria:

* Patient refuses study participation
* Severe renal failure
* Reduced life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for optimization of antihypertensive treatment to Luzerner Kantonsspital, Switzerland.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness and central hemodynamics | 3 months
  Non-invasive measurement of arterial stiffness and central hemodynamics with the Tensiomed Arteriograph device
Cognitive function | 3 months
  Measurement with Mini Mental State Exam and Verbal Recall Test

SECONDARY OUTCOMES:
Physical function | 3 months
  Measurement with gait speed, hand grip test and physical activity questionnaire
Orthostatic hypotension and falls | 3 months
  Measurement with blood pressure recordings and structured questionnaire
Renal failure | 3 months
  Creatinine measurement

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Study Chair — Luzerner Kantonsspital; Paul Erne, MD, Principal Investigator — Luzerner Kantonsspital; Andreas W Schoenenberger, MD, Principal Investigator — University hospital of Bern
Locations (1):
- Luzerner Kantonsspital, Lucerne, Canton of Lucerne, Switzerland